CLINICAL TRIAL: NCT03117036
Title: A Prospective Study for Patients With Lymphoid Malignancy at the Samsung Medical Center
Brief Title: Prospective Cohort Study for Lymphoma: Samsung Lymphoma Cohort Study III
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Samsung Genomic Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2016-11-040
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, Hodgkin
Keywords: lymphoma; cohort; serum; cell-free DNA
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma | interventions — Drug Therapy; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — serum and cell-free DNA from patients' peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lymphoma: Patients are diagnosed with aggressive lymphoma including Hodgkin and non-Hodgkin lymphoma. All patients should receive systemic chemotherapy. Newly diagnosed or relapsed/refractory patients can be enrolled.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Systemic chemotherapy with curative intent
  Other Names: Treatment

SUMMARY:
This prospective study enrolls patients who are diagnosed with aggressive lymphoma including Hodgkin and non-Hodgkin lymphomas. Enrolled patients will be treated according to our institution' treatment policy in clinical practice. The disease status including response to therapy and survival status will be regularly updated during the study period. Patients' serum and cell-free DNA will be collected and analyzed.

DETAILED DESCRIPTION:
The study population is aggressive lymphomas requiring systemic chemotherapy. Newly diagnosed or relapsed/refractory patients can be enrolled into the study. Patients can be treated according to the principle of routine care of our institute. The study process is as follows.

1. Registration after informed consent.
2. Laboratory and radiological evaluation after registration including collection of serum and cell-free DNA from patients' peripheral blood
3. Interim and final response evaluation including collection of serum and cell-free DNA from patients' peripheral blood
4. Regular monitoring disease status and update of survival status
5. Laboratory and radiological evaluation after relapse or progression including collection of serum and cell-free DNA from patients' peripheral blood

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed Hodgkin and non-Hodgkin lymphomas
2. 20 years
3. Patients requiring systemic chemotherapy with curative intent
4. Written informed consent

Exclusion Criteria:

1. Myeloid malignancy
2. Multiple myeloma
3. Patients do not require systemic chemotherapy with curative intent

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are diagnosed with aggressive lymphoma including Hodgkin and non-Hodgkin lymphoma. All patients should receive systemic chemotherapy. Newly diagnosed or relapsed/refractory patients can be enrolled
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Response rate | 3 months after chemotherapy
  response to chemotherapy

SECONDARY OUTCOMES:
Progression-free survival | 3 year
  Time to relapse/progression or any kinds of death
Overall survival | 3 year
  Time to any kinds of death
Biomarker | 3 year
  Development of biomarker predicting response and survival outcome

CONTACTS AND LOCATIONS:
Overall Officials: Seok Jin Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided